CLINICAL TRIAL: NCT05428540
Title: Influence of a Polyphenol-rich Supplement on Anthropometric, Biochemical and Inflammatory Parameters in Participants With Morbid Obesity
Brief Title: Polyphenol Supplementation and Morbid Obesity Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Raul Zamora Ros, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Polyphenols and morbid obesity
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Polyphenol-rich dietary supplement (3 capsules/day) + hypocaloric diet (1,200 kcal/day)
  Interventions: Dietary Supplement: Polyphenol-rich supplement
- Control group (Placebo Comparator): Placebo (3 capsules/day) + hypocaloric diet (1,200 kcal/day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Polyphenol-rich supplement — Polyphenol-rich capsules containing 1,200 mg of a combination of plant extracts rich in polyphenols. Frequency: 3 capsules a day. Duration: 12 weeks.
  Arms: Intervention group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
This parallel, double-blind, randomised controlled trial aims to assess the effect of a polyphenol-rich dietary supplement on obesity parameters, in combination with a hypocaloric diet, for adults with morbid obesity, bariatric surgery candidates.

Participants (n=40) will be randomly assigned to intervention group (IG) or control group (CG). Together with a regular hypocaloric diet (1,200 kcal/d), the IG will be given the supplement and the CG will be given a placebo. Both groups will take three capsules a day (400 mg per capsule, a total of 1,200 mg), distributed in three daily intakes (with meals). After 12 weeks and 3 visits (baseline visit, week 6 and week 12), pre and post intervention data and intervention versus placebo data will be analysed. Anthropometric and health parameters, dietary habits, lifestyle characteristics and physical activity will be assessed, and blood and urine samples will be collected in all three visits. Faecal samples will be collected at baseline and visit 3.

Results will provide evidence on the effects of a combination of polyphenols on several well-established obesity parameters and will unravel possible underlying mechanisms by metabolomic analyses and microbiota diversity.

DETAILED DESCRIPTION:
The main objective of this study is to assess the effect of a polyphenol-rich dietary supplement, along with a hypocaloric diet, on obesity parameters in participants with morbid obesity. Anthropometric, biochemical and inflammatory parameters, as well as different metabolic pathways and microbiota diversity will be assessed.

The estimated number of participants to include is 40. They will be patients with morbid obesity, referred to the Endocrinology and Nutrition Unit from Bellvitge University Hospital for a weight loss treatment, in many cases prior to a bariatric surgery. To estimate the sample size the following assumptions were made: same number of participants in each group; 10% variation in anthropometric and laboratory measurements; trial power of 0.85 and alfa error of 5%; estimated losses to follow-up: 15%.

The main component of the intervention is a polyphenol-rich dietary supplement administrated for 12 weeks. Lifestyle, dietary, physical activity data and blood and urine samples will be collected in three visits (baseline, week 6 and week 12); faecal samples will be collected in visits baseline and week 12. All participants will follow a hypocaloric diet and will be randomly assigned to either intervention group (IG) or control group (CG) after recruitment, following a simple randomisation procedure. The IG will take the supplement (3 capsules/day), whereas the CG will take a placebo (3 capsules/day).

This trial will be carried out following the ethical guidelines of the Declaration of Helsinki, the Principles of the Good Clinical Practice, under the existing legislation. Data collected will be kept strictly confidential. Any participant will have the right to access, rectification, cancellation and opposition over such data in accordance with the Organic Law 15/1999, Personal Data Protection. All information will be stored in a Data Collection Notebook, from which the database will be created.

All participants will be provided with an information sheet and will have to sign a consent form before the beginning of this trial. Any participant will be allowed to abandon the study for any reason: if requested; if the suspension is in the medical interest; if an incidence is presented as a consequence of the intervention, inacceptable or representing a threat to the participants' health; if the participant presents any breakthrough disease or other condition that, according to the principal investigator (PI), are relevant to suspend the intervention.

Data on medical history, lifestyle and sociodemographic characteristics will be collected through participants' clinical records and interviews at baseline. The standard hypocaloric diet (1200 kcal) that participants will have to follow for the entire 12 weeks of the study will be explained to each participant on the first visit.

On each visit participants will provide a 3-day food record, completed the three days preceding such visits. Qualified staff will collect data on dietary habits through a 24-hours dietary recall and will take anthropometric measurements, including height, weight, hip and waist circumference, body composition using an ergonomic measuring tape and a bioimpedance scan. Dietary and anthropometric assessment will be performed following the standard procedures from the Dietetic and Clinical Nutrition Unit from Bellvitge University Hospital.

Programari de Càlcul Nutricional Pro 1.0 Software, developed by University of Barcelona, will be used to assess dietary and nutritional intake. It includes a high-quality contrasted database which makes possible to calculate and analyse nutritional intake and body composition.

Phenol-Explorer database will be used to assess polyphenol intake. It is the first comprehensive database on polyphenol content in foods which takes into account food processing and cooking and contains more than 35,000 content values for 500 different polyphenols over 400 foods.

On each visit qualified staff will collect data on physical activity through a shortened version in Spanish of the Minnesota Leisure Time Physical Activity Questionnaire and will measure blood pressure through a semi-automated oscillometer.

Prior to each visit participants will need to fast for 12 hours as they will have blood samples taken. On each visit, 20ml of blood will be extracted from the antecubital vein and will be centrifuged and stored at -80ºC until used. Biochemical analyses will be performed by the Bellvitge University Hospital analysis laboratory. Blood tests will include rutinary hematology and biochemistry, and inflammatory parameters.

On each visit participants will have to 24-hour urine samples. Three aliquots (2 ml each) will be stored at -80ºC in the ultra-freezers of the Unit of Nutrition and Cancer, Institut d'Investigació Biomedica de Bellvitge (IDIBELL) (Barcelona, Spain). One aliquot will be used to measure cortisol in the clinical laboratory of the Bellvitge University Hospital. Another aliquot will be used to perform a metabolomic analysis by the Nutritional Biomarkers and Metabolomics group from the University of Barcelona. About ≈ 500 metabolites (e.g., polyphenols and microbiota metabolites, organic acids, energetic and protein metabolism compounds) will be quantified using ultra-high performance liquid chromatography coupled to tandem mass spectrometry. This will allow us to monitor metabolite alterations derived from the polyphenol-rich supplement and associate these changes with improvements in clinical and biochemical outcome measurements.

Participants will bring a faecal sample in the first and third visit. These samples will be analysed in future microbiota studies. They will be kept stored at -80ºC in the ultra-freezers of the Unit of Nutrition and Cancer, IDIBELL.

Statistical analysis plan: intention-to-treat and per-protocol analyses will be performed. The main variable to assess is body weight and body composition. Secondary variables include biochemical and inflammatory parameters, urine metabolites and microbiota. Pre and post data, and IG versus CG results will be compared using Student t-test for paired and for independent samples, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Presenting morbid obesity defined as BMI ≥ 40 kg/m2
* Referred to the Endocrinology and Nutrition Unit from Bellvitge University Hospital for a weight loss treatment

Exclusion Criteria:

* History of type I diabetes
* Endocrine disorders-derived obesity
* Acute metabolic complications
* Severe inflammatory process that might affect the inflammatory condition during the 4 weeks before inclusion
* Cardiovascular event during the 6 months before inclusion
* History of hepatopathy or alteration of hepatic function
* Pregnant, lactation period or willing to get pregnant in the 12 weeks after inclusion
* Recent history of neoplasia (< 5 years) except for skin cancer or melanoma
* Oral or IV line glucocorticoids during 14 consecutive days or more 3 months before inclusion
* Alcoholism, drug addiction or major psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Body weight | Visit 1 (baseline)
  Unit: Kilograms Measured with:bioimpedance scan
Body weight | Visit 2 (week 6)
  Unit: Kilograms Measured with:bioimpedance scan
Body weight | Visit 3 (week 12)
  Unit: Kilograms Measured with:bioimpedance scan

SECONDARY OUTCOMES:
Systolic blood pressure | Visit 1 (baseline)
  Unit: mmHg Measured with: oscillometer
Diastolic blood pressure | Visit 1 (baseline)
  Unit: mmHg Measured with: oscillometer
Systolic blood pressure | Visit 2 (week 6)
  Unit: mmHg Measured with: oscillometer
Diastolic blood pressure | Visit 2 (week 6)
  Unit: mmHg Measured with: oscillometer
Systolic blood pressure | Visit 3 (week 12)
  Unit: mmHg Measured with: oscillometer
Diastolic blood pressure | Visit 3 (week 12)
  Unit: mmHg Measured with: oscillometer
Dietary intake | Visit 1 (baseline)
  24-h dietary recall
Dietary intake | Visit 2 (week 6)
  24-h dietary recall
Dietary intake | Visit 3 (week 12)
  24-h dietary recall
Physical activity level | Visit 1 (baseline)
  Formula: metabolic energy turnover (MET) according to Ainsworth proposal (Compendium of Physical Activities, 2011) Unit: METS-minute/14 days
  Scale:
  <1250: sedentary 1250 to 2999: moderately active 3000-4999: active >=5000: very active
Physical activity level | Visit 2 (week 6)
  Formula: metabolic energy turnover (MET) according to Ainsworth proposal (Compendium of Physical Activities, 2011) Unit: METS-minute/14 days
  Scale:
  <1250: sedentary 1250 to 2999: moderately active 3000-4999: active >=5000: very active
Physical activity level | Visit 3 (week 12)
  Formula: metabolic energy turnover (MET) according to Ainsworth proposal (Compendium of Physical Activities, 2011) Unit: METS-minute/14 days
  Scale:
  <1250: sedentary 1250 to 2999: moderately active 3000-4999: active >=5000: very active
Alanine aminotransferase | Visit 1 (baseline)
  Measured through plasma concentrations:
  Unit: units/litre
Alanine aminotransferase | Visit 2 (week 6)
  Measured through plasma concentrations:
  Unit: units/litre
Alanine aminotransferase | Visit 3 (week 12)
  Measured through plasma concentrations:
  Unit: units/litre
Aspartate aminotransferase | Visit 1 (baseline)
  Measured through plasma concentrations Units: units/litre
Aspartate aminotransferase | Visit 2 (week 6)
  Measured through plasma concentrations Units: units/litre
Aspartate aminotransferase | Visit 3 (week 12)
  Measured through plasma concentrations Units: units/litre
Bilirrubin | Visit 1 (baseline)
  Measured through plasma concentrations Unit: mg/dl
Bilirrubin | Visit 2 (week 6)
  Measured through plasma concentrations Unit: mg/dl
Bilirrubin | Visit 3 (week 12)
  Measured through plasma concentrations Unit: mg/dl
Thyroid-stimulating hormone (TSH) | Visit 1 (baseline)
  Measured through plasma concentrations (mU/litre)
Thyroid-stimulating hormone (TSH) | Visit 2 (week 6)
  Measured through plasma concentrations (mU/litre)
Thyroid-stimulating hormone (TSH) | Visit 3 (week 12)
  Measured through plasma concentrations (mU/litre)
Thyroxine | Visit 1 (baseline)
  Measured through plasma concentrations (ng/dl)
Thyroxine | Visit 2 (week 6)
  Measured through plasma concentrations (ng/dl)
Thyroxine | Visit 3 (week 12)
  Measured through plasma concentrations (ng/dl)
Creatinin | Visit 1 (baseline)
  Measured through plasma concentrations (mg/dl)
Creatinin | Visit 2 (week 6)
  Measured through plasma concentrations (mg/dl)
Creatinin | Visit 3 (week 12)
  Measured through plasma concentrations (mg/dl)
Urea | Visit 1 (baseline)
  Measured through plasma concentrations (mg/dl)
Urea | Visit 2 (week 6)
  Measured through plasma concentrations (mg/dl)
Urea | Visit 3 (week 12)
  Measured through plasma concentrations (mg/dl)
Erithrocytes | Visit 1 (baseline)
  Plasma concentrations (cel/mcl)
Erithrocytes | Visit 2 (week 6)
  Plasma concentrations (cel/mcl)
Erithrocytes | Visit 3 (week 12)
  Plasma concentrations (cel/mcl)
Hemoglobin | Visit 1 (baseline)
  Plasma concentrations (g/dl)
Hemoglobin | Visit 2 (week 6)
  Plasma concentrations (g/dl)
Hemoglobin | Visit 3 (week 12)
  Plasma concentrations (g/dl)
Leucocytes | Visit 1 (baseline)
  Plasma concentrations (cel/mcl)
Leucocytes | Visit 2 (week 6)
  Plasma concentrations (cel/mcl)
Leucocytes | Visit 3 (week 12)
  Plasma concentrations (cel/mcl)
Total cholesterol | Visit 1 (baseline)
  Plasma concentrations (mg/dl)
Total cholesterol | Visit 2 (week 6)
  Plasma concentrations (mg/dl)
Total cholesterol | Visit 3 (week 12)
  Plasma concentrations (mg/dl)
LDL (low-density lipoprotein)-cholesterol | Visit 1 (baseline)
  Plasma concentrations (mg/dl)
LDL (low-density lipoprotein)-cholesterol | Visit 2 (week 6)
  Plasma concentrations (mg/dl)
LDL (low-density lipoprotein)-cholesterol | Visit 3 (week 12)
  Plasma concentrations (mg/dl)
HDL (high-density lipoprotein)-cholesterol | Visit 1 (baseline)
  Plasma concentrations (mg/dl)
HDL (high-density lipoprotein)-cholesterol | Visit 2 (week 6)
  Plasma concentrations (mg/dl)
HDL (high-density lipoprotein)-cholesterol | Visit 3 (week 12)
  Plasma concentrations (mg/dl)
Triglycerides | Visit 1 (baseline)
  Plasma concentrations (mg/dl)
Triglycerides | Visit 2 (week 6)
  Plasma concentrations (mg/dl)
Triglycerides | Visit 3 (week 12)
  Plasma concentrations (mg/dl)
Glucose | Visit 1 (baseline)
  Plasma concentrations (mg/dl)
Glucose | Visit 2 (week 6)
  Plasma concentrations (mg/dl)
Glucose | Visit 3 (week 12)
  Plasma concentrations (mg/dl)
Glycosylated hemoglobin | Visit 1 (baseline)
  Measured through plasma concentrations Unit: %
Glycosylated hemoglobin | Visit 2 (week 6)
  Measured through plasma concentrations Unit: %
Glycosylated hemoglobin | Visit 3 (week 12)
  Measured through plasma concentrations Unit: %
Insulin | Visit 1 (baseline)
  Measured through plasma concentrations Unit/ml
Insulin | Visit 2 (week 6)
  Measured through plasma concentrations Unit/ml
Insulin | Visit 3 (week 12)
  Measured through plasma concentrations Unit/ml
TNF-alpha receptor I | Visit 1 (baseline)
  Measured through plasma levels (pg/ml)
TNF-alpha receptor I | Visit 2 (week 6)
  Measured through plasma levels (pg/ml)
TNF-alpha receptor I | Visit 3 (week 12)
  Measured through plasma levels (pg/ml)
TNF-alpha receptor II | Visit 1 (baseline)
  Measured through plasma levels (pg/ml)
TNF-alpha receptor II | Visit 2 (week 6)
  Measured through plasma levels (pg/ml)
TNF-alpha receptor II | Visit 3 (week 12)
  Measured through plasma levels (pg/ml)
Interleukin-6 | Visit 1 (baseline)
  Measured through plasma levels (pg/ml)
Interleukin-6 | Visit 2 (week 6)
  Measured through plasma levels (pg/ml)
Interleukin-6 | Visit 3 (week 12)
  Measured through plasma levels (pg/ml)
Adiponectin | Visit 1 (baseline)
  Measured through plasma levels (ug/ml)
Adiponectin | Visit 2 (week 6)
  Measured through plasma levels (ug/ml)
Adiponectin | Visit 3 (week 12)
  Measured through plasma levels (ug/ml)
high sensitivity c-reactive protein | Visit 1 (baseline)
  Measured through plasma levels (mg/l)
high sensitivity c-reactive protein | Visit 2 (week 6)
  Measured through plasma levels (mg/l)
high sensitivity c-reactive protein | Visit 3 (week 12)
  Measured through plasma levels (mg/l)
Waist circumference | Visit 1 (baseline)
  Unit: centimetres Measured with: ergonomic measuring tape
Waist circumference | Visit 2 (week 6)
  Unit: centimetres Measured with: ergonomic measuring tape
Waist circumference | Visit 3 (week 12)
  Unit: centimetres Measured with: ergonomic measuring tape
Hip circumference | Visit 1 (baseline)
  Unit: centimetres Measured with: ergonomic measuring tape
Hip circumference | Visit 2 (week 6)
  Unit: centimetres Measured with: ergonomic measuring tape
Hip circumference | Visit 3 (week 12)
  Unit: centimetres Measured with: ergonomic measuring tape
Fat mass | Visit 1 (baseline)
  Unit: % Measured with: bioimpedance scan
Fat mass | Visit 2 (week 6)
  Unit: % Measured with: bioimpedance scan
Fat mass | Visit 3 (week 12)
  Unit: % Measured with: bioimpedance scan
Muscle mass | Visit 1 (baseline)
  Unit: % Measured with: bioimpedance scan
Muscle mass | Visit 2 (week 6)
  Unit: % Measured with: bioimpedance scan
Muscle mass | Visit 3 (week 12)
  Unit: % Measured with: bioimpedance scan

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain